Official Title of the study: Effect of breathing exercise on some physiological parameters, sleep quality and vitality in elderly.

**NCT number:** not yet have

**Date of the document:** January 1, 2019

## Informed Consent Form For Intervention Group

This study you attend is a scientific study and its name is "The Effect of Breathing Exercise on Some Physiological Parameters, Sleep Quality and Vitality in Elderly". The aim of the study is to determine the effect of breathing exercise on some physiological parameters, sleep quality and vitality in the elderly. Breathing exercises aim to get the maximal benefit from the lungs by focusing one's attention on breathing in, and out. Previous studies have demonstrated that breathing exercises increase lung volume, clear secretions, improve gas exchange, manage dyspnea and improve exercise capacity. Breathing exercises has no potential risk other than short-term dizziness.

In this study breathing exercises; between 18.02.2019 -09.05.2019, for 12 weeks, three days a week (Monday, Tuesday, Thursday), in groups of 5-6 people, between 10.00-15.30 hours, 30 minutes for each group at the same time of the day, will be applied. No special clothing or materials are needed during breathing exercises. The wind rose to be used during the exercise will be provided by the researcher. Before and after the application of respiratory exercise, with questionnaires and medical measurement tools, your lung functions, blood pressure, oxygen level in your blood, heart rate, sleep state, and body fitness will be checked. Assessment of lung functions will be done with a specialist physiotherapist. In addition, if any of the exclusion criteria of the study occurs during the exercise program, the researcher will be informed by the health unit and the elderly individual will be separated from the study. The study is carried out purely for research purposes. Participation is voluntary. Your information will only be used for scientific purposes.

Below is the exercise program to be implemented

- I. Pursed Lip Breathing Exercise (using the Wind rose)
- The individual is seated in a position where he feels comfortable and with clothes,
- First, breathe slowly through the nose,
- Lips contract like a whistle
- The wind rose is kept at the level of the mouth at a distance of 25 cm,
- The breath is discharged slowly and for a longer period of time (at least twice the breathing) by blowing from the shrunken lips to the wind rose,
- Power should be used to exhale,
- This process continues until the breath is interrupted,
- A break is taken for 30 seconds, then the procedure is repeated (Total 10 minutes)
- 2 minutes break

- II. Diaphragmatic breathing exercise
- The active hand is placed on the stomach and the other hand on the chest,
- Breathing slowly through your nose,
- The abdomen is filled with air and the hand rises,
- The rib cage should rise less than the abdomen,
- Then, breathing slowly through the mouth,
- 30 seconds break and the process is completed (10 minutes in total),
- 2 minutes break

## III. Cough exercise

- Then a deep breath is taken through the nose,
- After the chest is fully enlarged, mouth is exhaled,
- This process is repeated twice,
- Take a deep breath for the third time and hold it for 2 seconds,
- Then, two times, "huh huh" sound is made and the mouth is exhaled,
- 30 seconds break,
- Then this process is repeated (Total 10 minutes).

Thank you for your participation.

Gazi University Faculty of Health Sciences

Public Health Nursing Department

Researcher Researcher

Aysun ERDAL Prof. Dr. Naile B LGL

I have read the text of the above research, I know that I have the right to disagree or leave the trial at any stage of the trial. I voluntarily agree to participate in the study under these conditions

Date:

Signature:

## Informed Consent Form For Control Group

This study you attend is a scientific study and its name is "The Effect of Respiratory Exercise on Some Physiological Parameters, Sleep Quality and Fitness in the Elderly". The implementation of the research will be held between 18.02.2019 -09.05.2019. Within the scope of the research application, your lung function, blood pressure, oxygen level in your blood, heart rate, sleep state, and fitness of your body will be checked with surveys and medical measurement tools at the beginning and end of the study date. Apart from these measurements, any application that will continue normal daily life activities will not be carried out. No special clothing or material to be provided by the individual is required for the measurements. Evaluation of lung functions will be done in the presence of a specialist physiotherapist. These applications do not have any potential risk As a result of these measurements, you can have information about your lung function ,cadiological functions and sleep quality. The study is carried out purely for research purposes. Participation is voluntary. Your information will only be used for scientific purposes.

| 1 | hanl | k you | for you | r partici | pation. |
|---|------|-------|---------|-----------|---------|
|---|------|-------|---------|-----------|---------|

Gazi University Faculty of Health Sciences

Public Health Nursing Department

Researcher Researcher

Aysun ERDAL Prof. Dr. Naile B LGL

I have read the text of the above research, I know that I have the right to disagree or leave the trial at any stage of the trial. I voluntarily agree to participate in the study under these conditions

| Date: |
|-------|
|-------|

Signature: